CLINICAL TRIAL: NCT01784536
Title: Study Evaluating the Effects of a Single Oritavancin Infusion on Cytochrome P450 (CYP) 1A2, CYP2C9, CYP2C19, CYP2D6, CYP3A, N-Acetyltransferase-2, and Xanthine Oxidase Activities in Healthy Adults Using the Cooperstown 5 + 1 Cocktail
Brief Title: Open Label Study Evaluating the Effects of a Single Oritavancin Infusion on Cytochrome P450 in Healthy Volunteers
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-ORI-12-03
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oritavancin (Experimental): Single-Dose IV Oritavancin Diphosphate
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate

INTERVENTIONS:
Drug: Single-Dose IV Oritavancin Diphosphate — Oritavancin will be administered as a single IV infusion. The infusion will last approximately 3 hours.
  Other Names: Oritavancin Diphosphate

SUMMARY:
The purpose of this study is to examine the effects of oritavancin on the in vivo activities of CYP1A2, CYP2C9, CYP2C19, CYP2D6, CYP3A, NAT 2, and XO using a Cooperstown 5 + 1 cocktail in an open label, single arm manner.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent before study initiation.
* Healthy male or female adult between 18 and 45 years of age, inclusive.
* Body mass index (BMI) between 18 and 32 kg/m^2, inclusive.
* Nonsmoker for a 6-month period before Screening.
* In good health based upon results of medical history, physical examination, no clinically significant 12-lead ECG results, and laboratory test results.
* Agrees to avoid all medications (other than the study drugs) that may inhibit or induce hepatic microsomal enzymes during the study period, including prescription and nonprescription medications, vitamins, herbal supplements (including energy drinks), and nutraceuticals.
* Female subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use an acceptable nonhormonal method of contraception during all study phases.
* Agree to abstain from alcohol, caffeine-, and xanthine-containing products, all kind of energy drinks and the consumption of grapefruit juice and orange juice from 48 hours before study drug administration until completion of the follow-up visit.

Exclusion Criteria:

* Has acute or chronic respiratory disease.
* The use of nonprescription drugs during the 30-day period before screening.
* The use of any prescription drugs during the 3-month period before.
* Childbearing potential, a positive test result for urine or serum, human chorionic gonadotropin (hCG) at Screening.
* Positive serology result for hepatitis B surface antigen, hepatitis C virus antibody, or has known hepatitis B or C infection at screening.
* Positive serology result for human immunodeficiency virus (HIV) or has known immune deficiency disease at Screening.
* Requires anticoagulant monitoring with an activated partial thromboplastin time.
* Has an elevated international normalized ratio >1.3.
* Surgical or medical condition that could interfere with the administration of the study drug.
* Any condition that may affect drug absorption.
* Has a known intolerance to benzodiazepines, the active and/or inactive ingredients in caffeine, warfarin, vitamin K, omeprazole, or dextromethorphan.
* The use of any nicotine containing substance or nicotine replacement devices within 6 months before Screening.
* Has received an immunization during the 2-week period before screening.
* Has hemorrhagic tendencies or blood dyscrasias.
* Has poor venous access as determined by the investigator.
* Reports regular alcohol intake exceeding 1 drink/day within 1 month before screening.
* A poor metabolizer (based on medical history, if known) of CYP2D6, CYP2C9, or CYP2C19.
* Has participated in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days before enrollment.
* Excluded for any of the previous criteria may not be rescreened for participation at any time.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in the phenotyping measures of each probe drug in the absence and presence of oritavancin | Day 1 through Day 5

SECONDARY OUTCOMES:
Safety of probe drug administration and prolonged infusion of oritavancin as assessed by AEs/SAEs, clinical safety laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings | Day 1 through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States